CLINICAL TRIAL: NCT00497055
Title: Aripiprazole Treatment for Methamphetamine Dependence Among High-risk Individuals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: San Francisco Department of Public Health (Other Government)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Phillip Coffin, MD, MIA, Director of Substance Use Research, San Francisco Department of Public Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01DA022190-01 (NIH); 1R01DA022190-01 (NIH); 1R01DA023387-01 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Results first posted 2014-03-24 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-02

CONDITIONS: Substance Abuse; HIV Infections
Keywords: Methamphetamine; HIV; MSM; HIV Seronegativity
MeSH Terms: conditions — Substance-Related Disorders; HIV Infections | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aripiprazole (Experimental): Aripiprazole 5mg daily for week one. Aripiprazole 10mg daily for week two. Aripiprazole 20mg daily for weeks three through twelve.
  Interventions: Drug: Aripiprazole
- Placebo (Placebo Comparator): Placebo (for Aripiprazole) 5mg daily for week one. Placebo (for Aripiprazole) 10mg daily for week two. Placebo (for Aripiprazole) 20mg daily for weeks three through twelve.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole
  Other Names: Abilify
  Arms: Aripiprazole
Drug: Placebo — Sugar pill manufactured to mimic Aripiprazole gel caps.
  Arms: Placebo

SUMMARY:
Studies demonstrate that methamphetamine (meth) use is associated with high-risk sexual behavior among men who have sex with men (MSM), putting meth-using MSM at extraordinarily high risk for transmitting or acquiring HIV. This study is a randomized, double-blind, placebo-controlled trial of the medication aripiprazole for methamphetamine-using individuals, including MSM, and will assess efficacy, acceptability, tolerability, safety, and adherence to study medication.

DETAILED DESCRIPTION:
Population-based surveys estimate that the prevalence of methamphetamine use is 20 times higher among men who have sex with men (MSM) compared to the general population. Methamphetamine-associated sexual risk behavior is also a driving force in the MSM HIV epidemic: methamphetamine use has been associated with increased number of sexual partners, unprotected sex acts, sexually transmitted infections (STIs), and HIV acquisition. Despite these alarming data, relatively few interventions have been tested among methamphetamine-using MSM. Among heterosexual non-injection drug users, methamphetamine use has been associated with well characterized risks for HIV and STDs including increased numbers of sexual partners, less condom use than non-methamphetamine users, engaging in sex work, and self-reported history of STDs. In parallel with the continued testing of behavioral approaches, we believe the time has come to test the feasibility and acceptability of pharmacologic interventions to reduce methamphetamine use among high-risk individuals. Pharmacologic approaches to treating substance use have been successful in treating nicotine, alcohol, and heroin dependencies. Preliminary dosing studies demonstrate that aripiprazole (Abilify), an FDA-approved, well-tolerated antipsychotic and partial dopamine agonist, reduced the effects of methamphetamine in humans and exhibited a good safety profile. We propose to expand upon these promising results by conducting a randomized, double-blind, placebo-controlled pilot study of aripiprazole among sexually-active, methamphetamine-dependent individuals.

The specific aims of this study are:

1. To test the hypothesis that aripiprazole 20 mg daily will reduce methamphetamine use significantly more than placebo among methamphetamine-dependent individuals, as determined by the proportion of methamphetamine-negative urines and by self-report of methamphetamine use in the aripiprazole versus placebo group.
2. To measure the acceptability of aripiprazole and placebo among methamphetamine-dependent individuals, by determining (via electronic pill caps and self-report) medication adherence to aripiprazole and placebo.
3. To measure the safety and tolerability of aripiprazole and placebo among methamphetamine-dependent individuals, as determined by the number of adverse clinical events in the aripiprazole and placebo arms.

If promising, study results will be used to design larger, definitive clinical trials to determine the efficacy of aripiprazole in reducing methamphetamine use and corresponding methamphetamine-associated sexual risk among MSM. This pilot study is therefore designed to reflect the structure of such trials. We will enroll 90 sexually active, methamphetamine-dependent individuals who will be randomized 1:1 to receive aripiprazole (n=45) or placebo (n=45) for 12 weeks. Because we are testing a drug for a new indication in a new population, we will include extensive safety parameters, as done in prior studies of pharmacologic interventions among substance users. We will also include both urine testing and extensive behavioral risk assessments because we anticipate that future definitive efficacy trials will analyze both substance use and sexual risk behavior outcomes. Study participants will be seen at the San Francisco Department of Public Health AIDS Office where they will provide urines for drug testing and participate in substance use counseling. All participants will receive HIV risk-reduction counseling. Behavior will be assessed using standardized measures via audio computer-assisted self-interview (ACASI).

ELIGIBILITY:
A total of 90 high-risk individuals with methamphetamine dependence will be enrolled in the study. Subjects will be San Francisco Bay Area residents between 18-60 years of age and in good health. The project is designed specifically for those at high risk for HIV transmission or acquisition.

Inclusion Criteria:

1. HIV-negative by rapid test, or documentation of HIV infection with a laboratory result of a positive HIV test;
2. diagnosed with methamphetamine dependence as determined by SCID;
3. interested in stopping or reducing methamphetamine use;
4. at least one methamphetamine-positive urine during screening and run-in period;
5. no current acute illnesses requiring prolonged medical care;
6. no chronic illnesses that are likely to progress clinically during trial participation;
7. able and willing to provide informed consent and to be followed over trial period;
8. age 18-60 years;
9. baseline CBC, total protein, albumin, glucose, lipid panel, alk phos, creatinine, BUN, and electrolytes without clinically significant abnormalities as determined by investigator in conjunction with symptoms, physical exam, and medical history.
10. if sex assigned at birth was female and able to become pregnant: agrees to use birth control by any of the following methods - hormonal patch, pills, or injections; IUD; diaphragm; condoms; or abstinence.

Exclusion Criteria:

1. has a psychiatric disorder as assessed by SCID that in the opinion of evaluating clinician would make the study participation unsafe, or make adherence to study protocol untenable. Conditions include current major depression, current suicidal ideation, bipolar disorder, dementia, or acute psychosis;
2. taking psychotropic medication within the last 30 days, including aripiprazole;
3. known allergy to aripiprazole, or known adverse reaction to antipsychotics;
4. currently using or unwilling not to use phenylephrine or ephedrine-containing products for trial duration (can cause false positive urines for methamphetamine use);
5. current CD4 count < 200 cells/mm3;
6. using other medications known to interact with aripiprazole, including ketoconazole and carbamazepine;
7. measured moderate or severe liver disease (AST, ALT, and total bilirubin > 3 times normal) and/or any symptoms of current liver disease;
8. impaired renal function (creatinine clearance < 60 ml/min);
9. diabetes mellitis type I or type II, including cases controlled with diet alone;
10. Hypertension that is not well-controlled;
11. BMI ≥ 40; or BMI ≥ 35 with more than one of the following: age > 45, systolic blood pressure > 140 mm Hg, diastolic blood pressure > 90 mm Hg, known hyperlipidemia;
12. History of, or known active cardiovascular disease including: (a) Previous myocardial infarction (heart attack); (b) angina pectoris; (c) congestive heart failure; (d) valvular heart disease including mitral valve prolapse; (e) cardiomyopathy; (f) pericarditis; (g) stroke or transient ischemic attack; (h) chest pain or shortness of breath with activity (such as walking up stairs); (i) peripheral vascular disease or risk equivalent; (j) other heart conditions under the care of a doctor;
13. currently participating in another research study;
14. pregnant, breast-feeding, and/or positive pregnancy test at screening or enrollment visit;
15. any condition that, in the principal investigator's judgment, interferes with safe study participation or adherence to study procedures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2009-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip O Coffin, MD, MIA, Principal Investigator — Director of Substance Use Research, San Francisco Department of Public Health
Locations (1):
- San Francisco Department of Public Health, AIDS Office, San Francisco, California, United States

REFERENCES:
- [Result] Coffin PO, Santos GM, Das M, Santos DM, Huffaker S, Matheson T, Gasper J, Vittinghoff E, Colfax GN. Aripiprazole for the treatment of methamphetamine dependence: a randomized, double-blind, placebo-controlled trial. Addiction. 2013 Apr;108(4):751-61. doi: 10.1111/add.12073. Epub 2013 Jan 3. PMID 23186131

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aripiprazole | Placebo
Started | 45 | 45
Completed | 35 | 40
Not Completed | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Aripiprazole: aripiprazole daily for 3 months
- Placebo: placebo daily for 3 months
- Total: Total of all reporting groups
Arm/Group | Aripiprazole | Placebo | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 45 | 90
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (12.3) | 40 (8.9) | 38.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 39 | 40 | 79
Region of Enrollment [Number; unit: participants]
  United States | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: To Test the Hypothesis That Aripiprazole 20 mg Daily Will Reduce Methamphetamine Use Significantly More Than Placebo Among Methamphetamine-dependent Individuals.
Description: To test the hypothesis that aripiprazole 20 mg daily will reduce methamphetamine use significantly more than placebo among methamphetamine-dependent individuals, as determined by the proportion of methamphetamine-positive urines in the aripiprazole versus placebo group.
Time Frame: Final study visit at week 12
Measure: Number; unit: perc of positive urines at final visit
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 45 | 45
perc of positive urines at final visit | 44 | 40
Statistical Analysis 1: Comparison: Aripiprazole vs Placebo; Test type: Superiority or Other; p = .41, Generalized estimating equation; Risk Ratio (RR) = .88, 95% CI [.66 to 1.16]

2. Primary Outcome: To Measure the Acceptability of Aripiprazole and Placebo Among Methamphetamine-dependent Individuals, by Determining (Via Electronic Pill Caps [MEMS or Medication Event Monitoring System]) Medication Adherence to Aripiprazole and Placebo.
Description: To measure the acceptability of aripiprazole and placebo among methamphetamine-dependent individuals, by determining (via electronic pill caps [MEMS or Medication Event Monitoring System]) medication adherence to aripiprazole and placebo. (Percent adherence from MEMS is determined by 100* the number of days where MEMS registered an opening out of the number of days a dose was prescribed for each arm.)
Time Frame: Adherence as determined by MEMS (throughout study, up to 12 weeks)
Measure: Mean (Standard Deviation); unit: percent adherence from MEMS
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 45 | 45
percent adherence from MEMS | 46 (32) | 39 (27)
Statistical Analysis 1: Comparison: Aripiprazole vs Placebo; Test type: Superiority or Other; p = 0.31, Wilcoxon (Mann-Whitney)

3. Primary Outcome: To Measure the Safety and Tolerability of Aripiprazole and Placebo Among Methamphetamine-dependent Individuals, as Determined by the Number of Adverse Clinical Events in the Aripiprazole and Placebo Arms.
Time Frame: Total reported adverse events (throughout study, up to 12 weeks)
Measure: Number; unit: total reported adverse events
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 45 | 45
total reported adverse events | 156 | 144
Statistical Analysis 1: Comparison: Aripiprazole vs Placebo; Test type: Superiority or Other; p >= 0.99, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Aripiprazole | Placebo
Serious Adverse Events (participants affected / at risk) | 3/45 | 4/45
Other Adverse Events (participants affected / at risk) | 35/45 | 36/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole (N=45) | Placebo (N=45)
rhabdomyolysis (Renal and urinary disorders) | 1 | 0
subdural hematoma (Vascular disorders) | 0 | 1
metastatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
abscess (Skin and subcutaneous tissue disorders) | 0 | 2
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole (N=45) | Placebo (N=45)
Abrasions (Skin and subcutaneous tissue disorders) | 3 | 1
Akathisia (Nervous system disorders) | 12 | 2
Abscess (Skin and subcutaneous tissue disorders) | 1 | 4
Contusion (Skin and subcutaneous tissue disorders) | 1 | 4
Drowsiness (General disorders) | 6 | 0
Fatigue (General disorders) | 8 | 0
Hyperbilirubinemia (General disorders) | 3 | 4
Toothache (General disorders) | 3 | 4
Viral Syndrome (General disorders) | 1 | 3
Anxiety (Nervous system disorders) | 0 | 3
Depressed Mood (Psychiatric disorders) | 3 | 1
Gastroenteritis (Gastrointestinal disorders) | 1 | 4
Headache (Nervous system disorders) | 2 | 3
Hypernatremia (General disorders) | 4 | 0
Hypocalcemia (General disorders) | 3 | 2
Increased Alanine Transaminase (ALT) (General disorders) | 8 | 7
Increased Aspartate Transaminase (AST) (General disorders) | 6 | 4
Laceration (Skin and subcutaneous tissue disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 2 | 3
Restlessness (Nervous system disorders) | 4 | 1
Skin and soft tissue infection (Infections and infestations) | 3 | 5
Sleep Disturbance (Nervous system disorders) | 3 | 2
Sweats (General disorders) | 0 | 4
Upper Respiratory Infection (URI) (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Urinary Tract Infection (UTI) (Renal and urinary disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No